CLINICAL TRIAL: NCT05881187
Title: Analysis of the Outcomes of Photoactivated Chromophore for Keratitis Cross _linking for Treatment of Infectious Keratitis
Brief Title: Pack Cross Linking for Infectious Keratitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mariam Abdelmawgoud Mohamed, assistant lecteurer opthalmology department sohag univerisity hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pack cross linking
Record Dates: First submitted 2023-05-03; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Infectoius Keratitis
MeSH Terms: interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- groupA (control group) (Active Comparator): will include 20 eyes of 20 patients with infectious keratitis who will receive antimicrobial therapy.
  Interventions: Drug: Antibotice.g vigamox ED Antifungal e.g Dflucan
- group B (Active Comparator): will include 20 eyes of 20 patients with infectious keratitis who will undergo PACK accelerated cross-linking Protocol-1 (9 mW/cm2 for 10 minutes to achieve 5.4 J/cm2) followed by antimicrobial therapy
  Interventions: Drug: Riboflavin; Drug: Antibotice.g vigamox ED Antifungal e.g Dflucan; Device: pack cross linking
- group C (Active Comparator): will include 20 eyes of 20 patients with infectious keratitis who will undergo PACK accelerated crosslinking Protocol-2 (18 mW/cm2 for 7 minutes to achieve 7.2 J/cm2) followed by antimicrobial therapy
  Interventions: Drug: Riboflavin; Drug: Antibotice.g vigamox ED Antifungal e.g Dflucan; Device: pack cross linking

INTERVENTIONS:
Drug: Riboflavin — topical application of riboflavin followed by cross linking
  Arms: group B; group C
Drug: Antibotice.g vigamox ED Antifungal e.g Dflucan — topical application of antimicropial therapy
Device: pack cross linking — TOPICAL application of cross linking after application of Riboflavin TO TREAT INFECTIOUS KERATITIS
  Arms: group B; group C

SUMMARY:
The primary aim of this study is to investigate the efficiency of PACK_ CXL in treatment of infectious keratitis and analyze postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* are age ≥18 years, fungal, bacterial or mixed infectious keratitis, ulcer ≤ 4 mm in diameter and showing a maximum depth of 350 μm (as assessed by either optical coherence tomography (OCT))

Exclusion Criteria:

* age ≤18 years, viral infectious keratitis, non-infectiouskeratitis, melting corneal ulcers with impending perforation, corneal thickness < 400 μm (including the corneal epithelium) and systemic diseases or systemic surgery, single-eyed and immunosuppressed patients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
corneal THICKNESS | within 60 days
  decrease corneal THICKNESS USING ANTERIOR SEGMENT OPTICAL COHERENT TOPOGRAPHY

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Cabrera-Aguas M, Khoo P, Watson SL. Infectious keratitis: A review. Clin Exp Ophthalmol. 2022 Jul;50(5):543-562. doi: 10.1111/ceo.14113. Epub 2022 Jun 3. PMID 35610943
- [Background] Papaioannou L, Miligkos M, Papathanassiou M. Corneal Collagen Cross-Linking for Infectious Keratitis: A Systematic Review and Meta-Analysis. Cornea. 2016 Jan;35(1):62-71. doi: 10.1097/ICO.0000000000000644. PMID 26509768
- [Background] Tabibian D, Mazzotta C, Hafezi F. PACK-CXL: Corneal cross-linking in infectious keratitis. Eye Vis (Lond). 2016 Apr 19;3:11. doi: 10.1186/s40662-016-0042-x. eCollection 2016. PMID 27096139
- [Background] Kumar V, Lockerbie O, Keil SD, Ruane PH, Platz MS, Martin CB, Ravanat JL, Cadet J, Goodrich RP. Riboflavin and UV-light based pathogen reduction: extent and consequence of DNA damage at the molecular level. Photochem Photobiol. 2004 Jul-Aug;80:15-21. doi: 10.1562/2003-12-23-RA-036.1. PMID 15339215